CLINICAL TRIAL: NCT03666858
Title: An Observational, Single-Arm Study to Describe Pain Intensity, Pain Relief and Safety of Neosaldina in the Treatment of Tension-Type Headaches in Healthy Subjects
Brief Title: A Study to Describe Pain Intensity, Pain Relief and Safety of Neosaldina in the Treatment of Tension-type Headaches (TTH) in Healthy Participants
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Neosaldina-5001; U1111-1218-2357 (Registry Identifier: WHO)
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers; Tension-type Headache
Keywords: Drug Therapy
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neosaldina: Participants with episodic TTH and who have already been treated with Neosaldina will be included in the observation period of this study. During the observation period, participants will be administered with Neosaldina 2 tablets, orally in the beginning of the TTH episode, every 6 hours, and at maximum of 8 tablets per day, according to regular clinical practice of the physicians. The participants will be observed in this study from Day 1 until Day 45.

SUMMARY:
The purpose of this study is to describe pain relief in TTH with Neosaldina treatment.

DETAILED DESCRIPTION:
This is an observational, non-interventional and prospective study of healthy participants with episodic TTH who have already been treated with Neosaldina according to regular clinical practice. This study will assess the pain intensity and pain relief of TTH after the uptake of Neosaldina.

This study will enroll approximately 317 participants. All participants will be enrolled into one observational group:

• Neosaldina

Investigators will assess participants from the time of enrolment through the completion of observation period up to 6 months. Each participant will be assessed up to 45 days after first dose. The data will be collected from medical charts and during routine follow up visits. The data from participants will be collected through a self-administered questionnaire using a mobile phone. All the participants will be instructed to insert the data in an application, downloaded in their phone whenever they will have an episode of TTH and use Neosaldina.

This multi-center trial will be conducted in Brazil. The overall duration of observation period in this study is approximately 6 months. Participants will be contacted by telephone on Days 15 and 30 for a follow up and will make a final visit on Day 45.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of episodic TTH, as determined by the International Classification of Headache Disorders.
2. Healthy participants who was prescribed 2 tablets of Neosaldina for episodic TTH.
3. Receive treatment according to the Summary of Product Characteristics for Neosaldina.
4. Has access to a mobile phone with the ability to download the app with the study questionnaire.
5. Has at least 1 episode of TTH per month.

Exclusion Criteria:

1. Currently participates or plans to participate in an interventional clinical trial.
2. Has hypersensitivity or intolerance to dypirone (or pyrazolonic derivatives) or other components of the product formula.
3. Has history of migraine, cluster headaches, chronic TTH or any other type of primary headache other than episodic TTH.
4. Has suspected secondary headache.
5. Has serious comorbidities (hypertension, blood dyscrasias, malignant neoplasms, any type of hepatitis or kidney disease, disorders of the hematopoietic system, insufficient function of the bone marrow or certain metabolic diseases, such as hepatic porphyria or congenital deficiency of glucose-6-phosphate dehydrogenase) or taking any medications which might confound the pharmacological effects of the study drug (example immunosuppressive drugs, and beta blockers, anticonvulsivants, antidepressants) within 30 days before the start of study.
6. Women who may be pregnant or breastfeeding during the course of the study.
7. Has history of alcohol abuse or other drugs according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
8. Has mental incapacity, unwillingness or language barriers unable to understand the guidelines specified in this protocol.
9. Any other reason that, in the Investigator's opinion, makes the participant unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult participants with episodic TTH.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (5):
- Brazil (5):
  - Fundacao do ABC, Santo André, São Paulo
  - Universidade Metropolitana de Santos, Santos, São Paulo
  - Cemec Centro Multidisciplinar de Estudos Clinicos Ltda-Epp, São Bernardo do Campo, São Paulo
  - Sociedade Brasileira e Japonesa de Beneficencia Santa Cruz, São Paulo, São Paulo
  - Cepic- Centro Paulista de Investigacao Clinica E Servicos Medicos Ltda, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in Brazil from 20 December 2018 to 19 August 2019.
Pre-assignment Details: Healthy participants with episodic tension-type headache (TTH) who had at least 1 reported headache and Neosaldina intake in mobile phone application enrolled in Cohort 1. Participants from Cohort 1 who had pain intensity reported at 0 and 120 minutes after Neosaldina intake/0 pain before 120 minutes in first headache report enrolled in Cohort 2.
Groups:
- Cohort 1 (All Participants): Neosaldina: All healthy participants with at least one TTH episode and who were prescribed with 2 tablets of Neosaldina, orally, at maximum of 8 tablets per day for episodic TTH as per regular clinical practice were enrolled in this observational study on Day 1. Participants were instructed to insert the data in an application, downloaded onto mobile phone, whenever they had an episode of TTH and use Neosaldina. Participants were observed from Day 1 until Day 45. Data were also collected from medical charts and during the routine clinical appointment.
- Cohort 2 (Participants From Cohort 1): Neosaldina: All participants from Cohort 1 who reported pain intensity at 0 and 120 minutes after Neosaldina intake or reported 0 pain before 120 minutes in their first headache report and who were prescribed with 2 tablets of Neosaldina, orally, at maximum of 8 tablets per day for episodic TTH as per regular clinical practice were enrolled in this observational study on Day 1. Participants were instructed to insert the data in an application, downloaded onto mobile phone, whenever they had an episode of TTH and use Neosaldina. Participants were observed from Day 1 until Day 45. Data were also collected from medical charts and during the routine clinical appointment.
Period: Cohort 1
Arm/Group | Cohort 1 (All Participants): Neosaldina | Cohort 2 (Participants From Cohort 1): Neosaldina
Started | 216 (All participants with TTH who had reported at least one headache and Neosaldina intake.) | 0
Completed | 215 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Cohort 2
Arm/Group | Cohort 1 (All Participants): Neosaldina | Cohort 2 (Participants From Cohort 1): Neosaldina
Started | 0 | 138 (Cohort 1 participants with pain intensity at 0,120minutes after Neosaldina/0 pain before 120minutes.)
Completed | 0 | 137
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants with TTH who reported at least one headache episode and Neosaldina intake in the mobile phone application during the study.
Arm/Group | Cohort 1 (All Participants): Neosaldina
Number analyzed (Participants) | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.56 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172
  Male | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9
  Black or African American | 18
  White | 178
  Unknown or Not Reported | 11
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 216
Occupation [Count of Participants; unit: Participants]
  Employed | 130
  Employed and student | 52
  Homemaker | 13
  Student | 10
  Retired | 8
  Unemployed | 2
  Unknown | 1
Household Income [Count of Participants; unit: Participants]
  0.5 to 1 minimum wage | 4
  1 to 2 minimum wage | 15
  2 to 3 minimum wage | 49
  3 to 5 minimum wage | 43
  5 to 10 minimum wage | 45
  10 to 20 minimum wage | 43
  20 minimum wage | 7
  Not reported | 8
  No income | 1
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Cohort 2: Time-weighted Sum of Pain Intensity Difference From Baseline (0 Hour) to 2 Hours (SPID 0-2) Post-dose
Description: Sum of pain intensity difference (SPID) was calculated as time-weighted sum of the visual analogue scale (VAS) differences over 2 hour period. Pain intensity was measured by VAS which was an 11-point numerical rating scale, ranging from 0 (no pain) to 10 (very intense pain). Pain intensity difference (PID) was the difference between baseline pain intensity (prior to the dosing) and current pain intensity at assessment. Total possible score ranges from -720 (worst) to 120 (best) for SPID 0-2. A higher value in SPID indicated greater pain relief. This outcome was recorded at 15-minutes intervals for the first 60 minutes, followed by 30 minutes from 1 to 2 hours after Neosaldina administration.
Time Frame: Baseline (0 hour) up to 2 hours post-dose
Population: All participants from Cohort 1 with TTH who reported at least one headache episode and Neosaldina intake in the mobile phone application during the study and who reported pain intensity at 0 and 120 minutes after Neosaldina intake or reported 0 pain before 120 minutes in their first headache report, and with primary endpoint data available.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Cohort 2 (Participants From Cohort 1): Neosaldina
Number analyzed (Participants) | 138
units on a scale | -210 [-690 to 120]

2. Secondary Outcome: Cohorts 1 and 2: Percentage of Participants Who Achieved a Reduction of at Least 1 Point Pain in Intensity for Each Time Interval
Description: Pain intensity was measured by VAS which was an 11-point numerical rating scale, ranging from 0 (no pain) to 10 (very intense pain). Percentage of participants are reported who had no pain relief and who achieved a reduction of at least 1 point pain in intensity for each time interval.
Time Frame: 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, and 120 minutes
Population: All participants in Cohort(C)1 with TTH who had >=1 headache/Neosaldina intake in mobile application, from C1 in C2 who had pain intensity at 0, 120 minutes after Neosaldina intake,0 pain before 120 minutes in first headache report, with primary endpoint data. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (All Participants): Neosaldina | Cohort 2 (Participants From Cohort 1): Neosaldina
Number analyzed (Participants) | 152 | 138
percentage of participants
  At 15 minutes | 43.42 | 45.65
  At 30 minutes | 27.63 | 28.26
  At 45 minutes | 11.18 | 10.87
  At 60 minutes | 7.89 | 6.52
  At 90 minutes | 2.63 | 5.07
  At 120 minutes | 1.32 | 1.45
  No pain relief | 5.92 | 2.17

3. Secondary Outcome: Cohorts 1 and 2: Time to Achieve 50 Percent (%) of Pain Intensity Reduction
Description: Pain intensity was measured by VAS which was an 11-point numerical rating scale, ranging from 0 (no pain) to 10 (very intense pain).
Time Frame: Each episodic TTH (Day 1 up to Day 45)
Population: All participants in Cohort (C) 1 with TTH who had >=1 headache/Neosaldina intake in mobile application and from C1 in C2 who had pain intensity at 0, 120 minutes after Neosaldina intake/0 pain before 120 minutes in first headache report, and with primary endpoint data. Overall number analyzed are those who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cohort 1 (All Participants): Neosaldina | Cohort 2 (Participants From Cohort 1): Neosaldina
Number analyzed (Participants) | 125 | 132
minutes | 45.36 (26.63) | 51.36 (31.89)

4. Secondary Outcome: Cohorts 1 and 2: Time to First Perceptible Pain Relief (PR)
Description: The relief of pain intensity was assessed by the PID% in each time point. Pain intensity was measured by VAS which was an 11-point numerical rating scale, ranging from 0 (no pain) to 10 (very intense pain). PID was the difference between baseline pain intensity (prior to the dosing) and current pain intensity at assessment. Participants evaluated the time to first perceptible relief (confirmed by meaningful relief which was reduction of at least 1 point on pain intensity) according to the pain intensity reported at the time points 0, 15, 30, 45, 60, 90 and 120 minutes after Neosaldina administration.
Time Frame: Each episodic TTH (Day 1 to Day 45)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cohort 1 (All Participants): Neosaldina | Cohort 2 (Participants From Cohort 1): Neosaldina
Number analyzed (Participants) | 143 | 135
minutes | 30.31 (20.57) | 31.11 (22.34)

5. Secondary Outcome: Cohort 1: Mean Duration of PR for Participants With Second Neosaldina Intake
Description: Duration of PR was defined by the time of second intake of study medication.
Time Frame: Each episodic TTH (Day 1 up to Day 45)
Population: All participants with TTH who reported at least one headache episode and Neosaldina intake in the mobile phone application during the study. Here "overall number of participants" analyzed were those who had more than one headache in the same day and were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 (All Participants): Neosaldina
Number analyzed (Participants) | 6
hours | 5.16 (2.26)

6. Secondary Outcome: Cohorts 1 and 2: Number of Participants Categorized Based on Treatment Satisfaction According to Patient Global Assessments of Overall Satisfaction
Description: Overall satisfaction of participants was assessed by the participants based on Patient Global Assessment measured on a 5-point scale for TTH as: 0 (very satisfied); 1 (satisfied); 2 (indifferent); 3 (dissatisfied); 4 (very dissatisfied).
Time Frame: Day 45
Population: All participants in Cohort (C) 1 with TTH who had greater than or equal to (>=1) headache/Neosaldina intake in mobile application and from C1 in C2 who had pain intensity at 0, 120 minutes after Neosaldina intake/0 pain before 120 minutes in first headache report, and with primary endpoint data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (All Participants): Neosaldina | Cohort 2 (Participants From Cohort 1): Neosaldina
Number analyzed (Participants) | 216 | 138
Participants
  Very satisfied | 91 | 63
  Satisfied | 99 | 59
  Indifferent | 6 | 5
  Dissatisfied | 7 | 3
  Very dissatisfied | 2 | 1
  Unknown | 11 | 7

7. Secondary Outcome: Cohorts 1 and 2: Number of Participants Categorized Based on Treatment Satisfaction According to Physician Global Assessments of Overall Satisfaction
Description: Overall satisfaction of participants was assessed by the physicians based on Physician Global Assessment measured on a 5-point scale for TTH as: 0 (very satisfied); 1 (satisfied); 2 (indifferent); 3 (dissatisfied); 4 (very dissatisfied).
Time Frame: Day 45
Population: All participants in Cohort (C) 1 with TTH who had >=1 headache/Neosaldina intake in mobile application and from C1 in C2 who had pain intensity at 0, 120 minutes after Neosaldina intake/0 pain before 120 minutes in first headache report, and with primary endpoint data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (All Participants): Neosaldina | Cohort 2 (Participants From Cohort 1): Neosaldina
Number analyzed (Participants) | 216 | 138
Participants
  Very satisfied | 94 | 62
  Satisfied | 98 | 62
  Indifferent | 8 | 3
  Dissatisfied | 3 | 3
  Very dissatisfied | 2 | 1
  Unknown | 11 | 7

8. Secondary Outcome: Cohort 1: Number of Participants Who Experienced at Least One Adverse Event (AE) After Neosaldina Administration
Time Frame: Day 1 up to Day 45
Population: The safety analysis set included all participants with TTH who reported at least one headache episode and Neosaldina intake in the mobile phone application.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (All Participants): Neosaldina
Number analyzed (Participants) | 216
Participants | 6

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after Day 1 up to Day 45
Description: AEs are reported for the safety analysis set which included all participants who were enrolled in Cohort 1 with at least one headache report in the mobile phone application during the study. Incidence of adverse events was calculated based on the number of adverse events experienced divided by the total number of participants
Arm/Group | Cohort 1 (All Participants): Neosaldina
All-Cause Mortality (participants affected / at risk) | 0/216
Serious Adverse Events (participants affected / at risk) | 0/216
Other Adverse Events (participants affected / at risk) | 6/216
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (All Participants): Neosaldina (N=216)
Nausea (Gastrointestinal disorders) | 1
Sleepiness (Nervous system disorders) | 2
Lack of vitamin D (General disorders) | 1
Hypertension (Vascular disorders) | 1
Bacterial infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT03666858/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT03666858/SAP_001.pdf